CLINICAL TRIAL: NCT06719791
Title: The Safety and Efficacy Evaluation of Sirolomus as an Adjunctive Treatment for Focal Refractory Epilepsy: A Pilot Study
Brief Title: Sirolomus Adjuvant Treatment of Focal Refractory Epilepsy (SATFRE)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-259-002
Record Dates: First submitted 2024-12-01; First posted 2024-12-06 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Epilepsy, Drug Resistant
Keywords: Sirolomus; Focal Refractory Epilepsy; mTOR pathway
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open label single arm, drug sirolomus (Experimental): All subjects will receive the experimental drug
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Oral administration is given solely for the epilepsy seizure event. Dosage: The dosage is determined based on body surface area (BSA), with 0.5 mg per dose for BSA <1.2 m², 1 mg per dose for BSA 1.3-2.1 m², and 1.5 mg per dose for BSA >2.2 m².

SUMMARY:
The aim of this study is to evaluate the clinical efficacy of sirolimus as an adjunctive therapy for refractory epilepsy. The significance lies in addressing whether the mTOR inhibitor sirolimus has antiepileptic adjunctive effects for a broader range of patients with refractory epilepsy, with the hope of providing a new mTOR-targeted antiepileptic adjunctive medication regimen that is administered only during epileptic events and can be widely used for various types of refractory epilepsy.

DETAILED DESCRIPTION:
Previous research has shown that the mTOR pathway is involved in the "epilepsy memory" process. Associating the acute seizures of the mouse kainic acid epilepsy model with a specific odor stimulus can lead to specific induction of epileptic seizures by this odor stimulus two weeks later. After epileptic seizures induced by a specific odor stimulus, the expression of the memory-related molecule pmTOR in the mouse hippocampus changes in a time-dependent manner, indicating that the mTOR signaling pathway is involved in the reconsolidation process of epilepsy memory. Further intervention in the reconsolidation process of epilepsy memory with the mTOR inhibitor sirolimus (Rap) found that administering the drug within the memory consolidation window (5 min) could effectively intervene in the reinduction of epilepsy, while administering the drug outside the memory consolidation window (9 h) could not intervene. Professor Huang Zhuo's team validated the above experimental results using a conditioned epilepsy memory mouse model. Clinical experiments have found that administering the mTOR pathway inhibitor everolimus immediately after an epileptic seizure in patients can significantly reduce the interictal brain electrical activity, showing promising epilepsy treatment effects. However, this study only involved a single drug treatment, the treatment duration was short, and only the changes in epileptiform discharges after treatment with everolimus in epileptic patients were evaluated at the electrophysiological level, without evaluating the control efficacy on seizure symptoms in patients after repeated seizures with a sufficient course of treatment.

Therefore, inhibiting the mTOR signaling pathway within a specific time window by intervening in the reconsolidation of the current epileptic event holds promise as a new strategy to alleviate subsequent seizures. This strategy is expected to be applicable to a broader range of treatments for refractory epilepsy, and administering medication only during epileptic events is anticipated to achieve more efficient therapeutic effects.

Everolimus (sirolimus) is an inhibitor of the mammalian target of rapamycin (mTOR). In studies using animal models of tuberous sclerosis complex (TSC), mTOR inhibitors have been found to significantly reduce the frequency of epileptic seizures; furthermore, everolimus is currently undergoing phase III clinical trials as an adjunctive treatment for refractory epilepsy associated with TSC. Evidence from various animal models of epilepsy, including genetic epilepsy (such as in WAG/Rij rats) and acquired epilepsy (such as those induced by kainic acid or pilocarpine), also suggests the involvement of the mTOR signaling pathway in these forms of epilepsy and the broad inhibitory effects of mTOR inhibitors on epileptic seizures.

Based on the "epilepsy memory" mechanism, combining everolimus with a memory reconsolidation paradigm holds promise as an effective adjunctive treatment for refractory epilepsy. Evaluating its efficacy and safety not only helps establish its value in epilepsy treatment but also provides important guidance for clinical practice, crucial for the transition from basic research to clinical application.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age.
* Meet the 2017 International League Against Epilepsy (ILAE) diagnostic criteria for for focal seizures or focal seizures progressing to bilateral tonic-clonic seizures.
* Diagnosed with refractory epilepsy, having used at least two AEDs without effectiveness for 2 years. No drug interaction between current AEDs and sirolomus, and a stable dose for at least 12 weeks prior to enrollment.
* Seizure duration ≥1 minute, with accompanying sensory impairment.
* At least 6 focal seizures within the 12 weeks preceding enrollment.
* EEG or MRI/CT results within the past 2 years, confirming the diagnosis of focal epilepsy.
* The use of vagus nerve stimulation (VNS) and deep brain stimulation (DBS) is permitted, need to implant at least 5 months and stable for at least 12 weeks before enrollment.The parameters should keep unchanged until the end of the study.
* Informed consent signed.

Exclusion Criteria:

* Diagnosed with generalized or hereditary epilepsy with ion channel gene mutations
* Psychogenic non-epileptic seizures within 12 months;
* Treatable causes of epilepsy (such as metabolic disorders, toxicity, infections, space occupying lesions, or identified genetic abnormalities)
* Patients with only non-motor focal seizures, as classified by the 2017 ILAE.
* Seizure clusters within the 12 months.
* Tonic-clonic status epilepticus within12 months.
* Free of major medical illnesses including:
* Cerebrovascular events within the past 6 months, including cerebral infarction, cerebral hemorrhage, and transient ischemic attack, or those with progressive intracranial lesions.
* Severe uncontrolled diseases, such as immunodeficiency disorders, liver or kidney diseases, acute infections, or advanced-stage tumors.
* Severe cardiovascular or peripheral vascular diseases, such as those classified as NYHA Class III-IV, or those with malignant arrhythmias (e.g., Long QT syndrome, Brugada syndrome, and conduction block), or any other clinically significant electrocardiogram abnormalities, or who have had a myocardial infarction within the past 3 months before screening
* Participants with a history of medical conditions or surgeries that, in the investigator's judgment, could affect the absorption, distribution, or metabolism of the study drug (e.g., active peptic ulcers, ulcerative colitis, Crohn's disease, or bowel obstruction) or those with difficulty swallowing.
* Participants with any medical condition, mental health status, cognitive impairment, or intellectual disability that the investigator believes could increase the risk to the participant or interfere with their ability to participate in the clinical trial.
* Severe allergic reactions to any component of sirolimus, or have hypersensitivity.
* Participants meeting any of the following laboratory criteria: alanine aminotransferase (ALT) >2× upper limit of normal (ULN), aspartate aminotransferase (AST) >2× ULN, alkaline phosphatase (ALP) >2× ULN, platelet count <80×10^9/L, neutrophil count <1.8×10^9/L, or creatinine clearance (CLcr) <30 mL/min (calculated by the Cockcroft-Gault formula).
* In the period of pregnancy, childbirth, lactation.
* Alcohol abuse or drug misuse within 2 years prior to medication.
* Participation in another clinical study within 3 months;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Seizure Frequency Per 28 Days | assessed per 28 days during the treatment.
  Percent change in 28-day frequency of seizures during the 40 week treatment and follow-up period relative to baseline
50% Seizure Responder Rate | short-term treatment period (ending at 3 months); long-term follow-up period (ending at 12 months).
  The proportion of patients with a ≥ 50% reduction from Baseline in seizure frequency.

SECONDARY OUTCOMES:
Seizure Severity | Baseline observation period; short-term treatment period (ending at 3 months); long-term follow-up period (ending at 12 months).
  The percent change from baseline in seizure severity evaluated by Liverpool seizure severity scale (LSSS) .
Life quality evaluation | Baseline observation period; short-term treatment period (ending at 3 months); long-term follow-up period (ending at 12 months).
  Percentage change from baseline in Quality of Life in Epilepsy-31 inventory (QOLIE-31) score.
Adverse Events | through study completion, 12 months.
  Rate of adverse events which were judged to be study-related throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing; Zhuo Huang, PhD, Principal Investigator — Peking University School of Pharmaceutical Sciences
Locations (1):
- Xuanwu Hospital, Beijing, China